CLINICAL TRIAL: NCT06480968
Title: Safety and Tolerability of CTH120, First-in-human Phase I Study Encompassing Three Parts: Single and Multiple Ascending Doses and Potential Food Interaction
Brief Title: CTH120 First-in-Human Study: Single and Multiple Ascending Doses and Potential Food Interaction
Acronym: FIH-CTH120
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Connecta Therapeutics, S.L. (Industry)
Collaborators: Hospital del Mar Research Institute (IMIM) (Other); Adknoma Health Research (Industry); Ministry of Science and Innovation, Spain (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTH-CTH120-FIH-01; 2022-502209-13-01 (Other: EU CT Number)
Record Dates: First submitted 2023-07-27; First posted 2024-07-01 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Fragile X Syndrome
Keywords: Fragile X Syndrome; FXS; Fragile X; Neurodevelopmental Disorders; Central Nervous System Diseases; Intellectual Disability; Neurobehavioral Manifestations; Genetic Diseases, X-Linked; Congenital Abnormalities; Orphan Diseases; Rare Diseases
MeSH Terms: conditions — Fragile X Syndrome; Neurodevelopmental Disorders; Central Nervous System Diseases; Intellectual Disability; Neurobehavioral Manifestations; Genetic Diseases, X-Linked; Congenital Abnormalities; Rare Diseases

STUDY DESIGN:
Intervention Model Description: FIH-CTH120-SAD: Prospective, monocentre, double-blind, randomized, placebo-controlled, subsequent-group, Phase I investigation to assess the safety, tolerability and pharmacokinetics of CTH120 administered orally in single ascending doses.
  FIH-CTH120-MAD: Prospective, monocentre, double-blind, randomized, placebo-controlled, subsequent-groups, Phase I investigation to assess the safety, tolerability and pharmacokinetics of CTH120 administered orally in multiple ascending doses.
  FIH-CTH120-FI: Prospective, open-label single dose, two-condition (fed versus fasting), two sequences, crossover Phase I investigation to assess the effects of food on the bioavailability of CTH120.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: FIH-CTH120-SAD and FIH-CTH120-MAD: double-blind, placebo-controlled trial preventing the knowledge of the study drug allocation. Thus, all trial stakeholders but the Pharmacy personnel will be blinded throughout the trial including the Sponsor personnel, the participating subjects, the study team at the investigational site, including the person administering the study drugs to the subject as well as the CRO personnel involved in the data management and statistical analysis.
  FIH-CTH120-FI: open-label study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CTH120 (Experimental): Hard capsules of two strengths, 10 mg and 75 mg of CTH120 to be administered with 200 mL of water. CTH120 will be supplied by CONNECTA Therapeutics. Within each dose cohort group subjects (n=8) will be randomly assigned to the CTH120 dose or to the matching placebo in a 6 to 2 randomization ratio (placebo=2 and CTH120=6 per dose).
  Interventions: Drug: CTH120
- Placebo (Placebo Comparator): Hard capsules of placebo to be administered with 200 mL of water. Placebo will be supplied by CONNECTA Therapeutics. Within each dose cohort group subjects (n=8) will be randomly assigned to the CTH120 dose or to the matching placebo in a 6 to 2 randomization ratio (placebo=2 and CTH120=6 per dose).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: CTH120 — FIH-CTH120-SAD: Each independent cohort of 8 subjects (placebo=2 and CTH120=6 per dose) will receive a single administration of CTH120 or placebo. Four consecutive dose levels (20 mg/day, 40 mg/day, 85 mg/day and 160 mg/day) are planned. If no significant clinical adverse events are observed in the FIH-CTH120-SAD phase, an additional 5th cohort will be recruited to conduct the 5th dose level.
  FIH-CTH120-MAD: Each independent cohort of 8 subjects (placebo=2 and CTH120=6 per dose) will receive a daily administration of CTH120 or placebo for 7 days. Three consecutive dose levels are planned. The starting dose will be confirmed following the observed results of FIH-CTH120-SAD.
  FIH-CTH120-FI: One dosage of CTH120 will be assessed in 12 healthy male and female subjects in two conditions (Fed and Fasting). Subjects will be randomly assigned to 2 sequences: 6 subjects in a sequence "fed then fasting condition", 6 subjects in the reverse sequence ("fasting, then fed condition").
  Arms: CTH120
Other: Placebo — FIH-CTH120-SAD: Each independent cohort of 8 subjects (placebo=2 and CTH120=6 per dose) will receive a single administration of CTH120 or placebo. Four consecutive dose levels (20 mg/day, 40 mg/day, 85 mg/day and 160 mg/day) are planned. If no significant clinical adverse events are observed in the FIH-CTH120-SAD phase, an additional 5th cohort will be recruited to conduct the 5th dose level.
  FIH-CTH120-MAD: Each independent cohort of 8 subjects (placebo=2 and CTH120=6 per dose) will receive a daily administration of CTH120 or placebo for 7 days. Three consecutive dose levels are planned. The starting dose will be confirmed following the observed results of FIH-CTH120-SAD.
  Arms: Placebo

SUMMARY:
The purpose of this First-in-Human Phase I study is to investigate the safety, tolerability and pharmacokinetics of CTH120 in adult healthy volunteers.

DETAILED DESCRIPTION:
This trial is divided in three parts: FIH-CTH120-SAD (Single Ascending Doses), FIH-CTH120-MAD (Multiple Ascending Doses) and FIH-CTH120-FI (Food Interaction). FIH-CTH120-SAD will start first. The start of FIH-CTH120-MAD will await the results of at least three cohorts from the FIH-CTH120-SAD study before initiated. The starting dose of the FIH-CTH120-MAD will have been shown to be well tolerated in FIH-CTH120-SAD. FIH-CTH120-FI will be the last to start.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects: As the effect of the study drug on sperm is still unknown, male subjects should refrain from donating sperm or plan a pregnancy with their partner throughout the study and after 90 days after the trial and must report immediately to the study doctor if its partner becomes pregnant during the study and during 90 days after the study. The male subject will have to use double- barrier contraceptive methods: male condoms and spermicide.
* Healthy female subjects of non-child-bearing potential: females may be accepted if they are documented to be surgically sterile i.e., hysterectomy, tubal ligation or post-menopausal with a negative pregnancy test.
* Age ≥ 18 and ≤ 55 years.
* Weight ≥ 50 kg and ≤ 100 kg.
* Body mass index (BMI) ≥ 18 and ≤ 30.
* Negative serum pregnancy test (women only).
* Non-smoking.
* No history of or ongoing clinically relevant diseases or conditions.
* No clinically relevant findings in physical examination, vital signs (blood pressure, heart rate and body temperature), ECG and safety laboratory parameters that should be within normal ranges or considered as non-clinically relevant by the investigator.
* Able/willing to accept restrictions regarding diet, physical exercise, and consumption of alcohol and/or xanthine containing items during the duration of the trial including when out of CRU.
* Able to read Spanish or Catalan and adhere to study requirements.
* Not under any administrative or legal supervision.
* Signed informed consent prior to any study-mandated procedure.

Exclusion Criteria:

* Women of child-bearing potential.
* Life-time substance use disorders (SUD) according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-5).
* Recreational use of drugs of abuse within the last month prior to study drug administration (verified by hair testing).
* Positive blood or urine test for drugs of abuse or alcohol breath test prior to study drug administration.
* Life-time history of mental diseases.
* History of anxiety or depression not completely recovered within 12 months prior to study drug administration, as assessed by the Dual Diagnosis Screening Interview (DDSI).
* Clinically relevant cognitive impairment preventing the administration of the psychometric tests.
* Any other clinically relevant disease or condition that in the judgment of the investigator might interfere with the subject's ability to comply with study procedures or requirements and/or bias the interpretation of the study results and/or jeopardize the subject's safety.
* Ongoing gastrointestinal diseases or history of gastrointestinal surgery affecting absorption.
* Subjects with a clinically significant disease within one month prior to study drug administration.
* Any clinically relevant findings in physical examination, vital signs, ECG and safety laboratory parameters.
* A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms).
* A history of additional risk factors for TdP (e.g., heart failure, hypokalaemia, family history of Long QT Syndrome).
* The use of concomitant medications that prolong the QT/QTc interval.
* Positive hepatitis or HIV test.
* Known hypersensitivity to drug or drug excipients.
* Use of drugs known to induce or inhibit hepatic drug metabolism within one month prior to study administration or during the study and use of citrus juice during the study.
* Any prescription or over-the-counter (OTC) product including herbal, homeopathic, vitamins, minerals and nutritional supplements within 2 weeks (or more, considering the elimination half-life of the product) prior to study drug administration.
* Donation of blood or plasma within one month prior to study drug administration or transfusion of blood or plasma for medical/surgical reasons or intention to donate blood or plasma within one month after study drug administration.
* History of inadequate venous access and/or experience of difficulty donating blood.
* Not able/not willing to accept restrictions regarding diet, physical exercise, and consumption of alcohol and/or xanthine containing items when out of CRU.
* Subject included in a clinical study within 3 months prior to study drug administration.
* Subject already included in other parts of this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2023-06-23 (Actual); Primary Completion 2024-11-11 (Actual); Study Completion 2024-11-11 (Actual)

PRIMARY OUTCOMES:
Treatment-emergent adverse events (TEAEs). | From Day 1 to End-of-study: EOS will be on Day 8 (± 1 day) for FIH-CTH120-SAD and on Day 15 (+ 2 days) for FIH-CTH120-MAD
  Primary Safety and Tolerability endpoint for FIH-CTH120-SAD and FIH-CTH120-MAD (Not applicable for FIH-CTH120-FI).
  • AEs will be described in terms of result, frequency, intensity, medical decision, relation with study drug, as well as treatment received and subject retirement, duration, and time elapsed. AEs will also be listed and coded using the MedDRA Dictionary (version 26.0) for the term's codification.
Treatment-emergent potentially clinically significant abnormalities (PSCAs) in blood pressure (mmHg) | From Day 1 to End-of-study (EOS): on Day 8 (± 1 day) for FIH-CTH120-SAD, and on Day 15 (+ 2 days) for FIH-CTH120-MAD
  Primary Safety and Tolerability endpoint for FIH-CTH120-SAD and FIH-CTH120-MAD (Not applicable for FIH-CTH120-FI).
  • Blood pressure (mmHg) will be measured in the supine position following a 5 min rest.
Treatment-emergent potentially clinically significant abnormalities (PSCAs) in pulse rate (bpm) | From Day 1 to End-of-study (EOS): on Day 8 (± 1 day) for FIH-CTH120-SAD, and on Day 15 (+ 2 days) for FIH-CTH120-MAD
  Primary Safety and Tolerability endpoint for FIH-CTH120-SAD and FIH-CTH120-MAD (Not applicable for FIH-CTH120-FI).
  • Pulse rate (bpm) will be measured in the supine position following a 5 min rest.
Treatment-emergent potentially clinically significant abnormalities (PSCAs) in oral body temperature (ºC) | From Day 1 to End-of-study (EOS): on Day 8 (± 1 day) for FIH-CTH120-SAD, and on Day 15 (+ 2 days) for FIH-CTH120-MAD
  Primary Safety and Tolerability endpoint for FIH-CTH120-SAD and FIH-CTH120-MAD (Not applicable for FIH-CTH120-FI).
  • Oral body temperature (ºC) will be measured using an automated vital sign monitor device.
Treatment-emergent potentially clinically significant abnormalities (PSCAs) in electrocardiogram (ECG) values: normal sinus rhythm (NSR) | From Day 1 to End-of-study (EOS): on Day 8 (± 1 day) for FIH-CTH120-SAD, and on Day 15 (+ 2 days) for FIH-CTH120-MAD
  Primary Safety and Tolerability endpoints for FIH-CTH120-SAD and FIH-CTH120-MAD (Not applicable for FIH-CTH120-FI)
  • Computerized 12-lead electrocardiogram (ECG) recordings will be obtained. Each lead shall be recorded for at least 3 beats at a speed of 25 mm/s. Triplicate recordings will be made at the time points evaluated. The following parameter will be recorded: normal sinus rhythm (NSR).
Treatment-emergent potentially clinically significant abnormalities (PSCAs) in electrocardiogram (ECG) values: heart rate (bpm) | From Day 1 to End-of-study (EOS): on Day 8 (± 1 day) for FIH-CTH120-SAD, and on Day 15 (+ 2 days) for FIH-CTH120-MAD
  Primary Safety and Tolerability endpoints for FIH-CTH120-SAD and FIH-CTH120-MAD (Not applicable for FIH-CTH120-FI)
  • Computerized 12-lead electrocardiogram (ECG) recordings will be obtained. Each lead shall be recorded for at least 3 beats at a speed of 25 mm/s. Triplicate recordings will be made at the time points evaluated. The following parameter will be recorded: heart rate (bpm).
Treatment-emergent potentially clinically significant abnormalities (PSCAs) in electrocardiogram (ECG) values: PR interval (ms) | From Day 1 to End-of-study (EOS): on Day 8 (± 1 day) for FIH-CTH120-SAD, and on Day 15 (+ 2 days) for FIH-CTH120-MAD
  Primary Safety and Tolerability endpoints for FIH-CTH120-SAD and FIH-CTH120-MAD (Not applicable for FIH-CTH120-FI)
  • Computerized 12-lead electrocardiogram (ECG) recordings will be obtained. Each lead shall be recorded for at least 3 beats at a speed of 25 mm/s. Triplicate recordings will be made at the time points evaluated. The following parameter will be recorded: PR interval (ms).
Treatment-emergent potentially clinically significant abnormalities (PSCAs) in electrocardiogram (ECG) values: QRS duration (ms) | From Day 1 to End-of-study (EOS): on Day 8 (± 1 day) for FIH-CTH120-SAD, and on Day 15 (+ 2 days) for FIH-CTH120-MAD
  Primary Safety and Tolerability endpoints for FIH-CTH120-SAD and FIH-CTH120-MAD (Not applicable for FIH-CTH120-FI)
  • Computerized 12-lead electrocardiogram (ECG) recordings will be obtained. Each lead shall be recorded for at least 3 beats at a speed of 25 mm/s.Triplicate recordings will be made at the time points evaluated. The following parameter will be recorded: QRS duration (ms).
Treatment-emergent potentially clinically significant abnormalities (PSCAs) in electrocardiogram (ECG) values: QT (ms) | From Day 1 to End-of-study (EOS): on Day 8 (± 1 day) for FIH-CTH120-SAD, and on Day 15 (+ 2 days) for FIH-CTH120-MAD
  Primary Safety and Tolerability endpoints for FIH-CTH120-SAD and FIH-CTH120-MAD (Not applicable for FIH-CTH120-FI)
  • Computerized 12-lead electrocardiogram (ECG) recordings will be obtained. Each lead shall be recorded for at least 3 beats at a speed of 25 mm/s.Triplicate recordings will be made at the time points evaluated. The following parameter will be recorded: QT (ms).
Treatment-emergent potentially clinically significant abnormalities (PSCAs) in electrocardiogram (ECG) values: QTcF (ms) | From Day 1 to End-of-study (EOS): on Day 8 (± 1 day) for FIH-CTH120-SAD, and on Day 15 (+ 2 days) for FIH-CTH120-MAD
  Primary Safety and Tolerability endpoints for FIH-CTH120-SAD and FIH-CTH120-MAD (Not applicable for FIH-CTH120-FI)
  • Computerized 12-lead electrocardiogram (ECG) recordings will be obtained. Each lead shall be recorded for at least 3 beats at a speed of 25 mm/s.Triplicate recordings will be made at the time points evaluated. The following parameter will be recorded: QTcF (ms).
Treatment-emergent potentially clinically significant abnormalities (PSCAs) in safety laboratory parameters: haematology | From Day 1 to End-of-study (EOS): on Day 8 (± 1 day) for FIH-CTH120-SAD, and on Day 15 (+ 2 days) for FIH-CTH120-MAD
  Primary Safety and Tolerability endpoints for FIH-CTH120-SAD and FIH-CTH120-MAD (Not applicable for FIH-CTH120-FI). The following tests will be performed:
  • Haematology: complete blood count (complete blood count [CBC]; including haemoglobin, haematocrit, red blood cell [RBC], white blood cell (WBC), platelet count, and percent and absolute differential count (neutrophils, lymphocytes, eosinophils, monocytes, basophils, and other cells).
Treatment-emergent potentially clinically significant abnormalities (PSCAs) in safety laboratory parameters: serum chemistry | From Day 1 to End-of-study (EOS): on Day 8 (± 1 day) for FIH-CTH120-SAD, and on Day 15 (+ 2 days) for FIH-CTH120-MAD
  Primary Safety and Tolerability endpoints for FIH-CTH120-SAD and FIH-CTH120-MAD (Not applicable for FIH-CTH120-FI). The following tests will be performed:
  • Serum chemistry: sodium, potassium, chloride, non-fasting glucose, urea, creatinine, calcium, phosphate, magnesium, total and direct bilirubin, total protein, albumin, ALT, AST, ALP, lactate dehydrogenase.
Treatment-emergent potentially clinically significant abnormalities (PSCAs) in safety laboratory parameters: coagulation | From Day 1 to End-of-study (EOS): on Day 8 (± 1 day) for FIH-CTH120-SAD, and on Day 15 (+ 2 days) for FIH-CTH120-MAD
  Primary Safety and Tolerability endpoints for FIH-CTH120-SAD and FIH-CTH120-MAD (Not applicable for FIH-CTH120-FI). The following tests will be performed:
  • Coagulation parameters: activated partial thromboplastin time (aPTT), PT and INR.
Treatment-emergent potentially clinically significant abnormalities (PSCAs) in safety laboratory parameters: urinalysis | From Day 1 to End-of-study (EOS): on Day 8 (± 1 day) for FIH-CTH120-SAD, and on Day 15 (+ 2 days) for FIH-CTH120-MAD
  Primary Safety and Tolerability endpoints for FIH-CTH120-SAD and FIH-CTH120-MAD (Not applicable for FIH-CTH120-FI). The following tests will be performed:
  • Urinalysis parameters:
  * Macroscopic examination: specific gravity, pH, protein, glucose, ketones, blood, bilirubin, leukocyte, urobilinogen, and nitrite.
  * Microscopic examination: RBCs, WBCs, epithelial cells, casts, crystals, bacteria, and yeast.
Psychometric tests: Hospital Anxiety/Depression rating Scale (HADS) | FIH-CTH120-SAD: on Day -1 and Day 2; FIH-CTH120-MAD: on Day -1, Day 1, and Day 7
  Primary Safety and Tolerability endpoints for FIH-CTH120-SAD and FIH-CTH120-MAD (Not applicable for FIH-CTH120-FI).
  • HADS: Self-reported questionnaire used to detect depression and anxiety. It consists of 14 items (7 related to depression and 7 to anxiety) scored using a 4-point Likert scale (each item ranging from 0 to 3). Two scores are generated one for depression and one for anxiety each score ranging from 0 to 21. Higher scores indicate greater levels of anxiety or depression. Both scores can be categorized into: Normality (0-7); Probable case of anxiety or depression (8-10); Case of anxiety or depression (11-21).
Psychometric tests:Immediate Mood Scaler (IMS). | FIH-CTH120-SAD: on Day -1 and Day 2; FIH-CTH120-MAD: on Day -1, Day 1, and Day 7
  Primary Safety and Tolerability endpoints for FIH-CTH120-SAD and FIH-CTH120-MAD (Not applicable for FIH-CTH120-FI).
  • IMS: The IMS is a tool to remotely and quickly track mood changes related to depression and anxiety in the moment. It consists of 22 items, scored between 1 and 7. The total score for this scale is the sum of the scores on all 22 items: ranging from 22 to 154. Lower scores reflect more negative mood states.
Area under the concentration-time curve (AUC0-24h, AUC0-t, AUC0-∞) after fed and fasting conditions. | FIH-CTH120-FI: AUC0-24h on Day 1; AUC0-t, AUC0-∞ where t is the last or the latest timepoint observed
  Primary Pharmacokinetic endpoint for FIH-CTH120-FI (Not applicable for FIH-CTH120-SAD and FIH-CTH120-MAD).
  • Plasma PK parameter calculated using a non-compartmental model: AUC0-24h (h * ng/mL), AUC0-t (h * ng/mL) AUC0-∞ (h * ng/mL).
Observed maximum concentration (Cmax) after fed and fasting conditions. | FIH-CTH120-FI: On Day 1 of Period 1, and on Day 14/21/25 of Period 2
  Primary Pharmacokinetic endpoint for FIH-CTH120-FI (Not applicable for FIH-CTH120-SAD and FIH-CTH120-MAD)
  • Plasma PK parameter calculated using a non-compartmental model: Cmax (ng/mL).
Time to observed maximum concentration (tmax) after fed and fasting conditions. | FIH-CTH120-FI: On Day 1 of Period 1, and on Day 14/21/25 of Period 2
  Primary Pharmacokinetic endpoint for FIH-CTH120-FI (Not applicable for FIH-CTH120-SAD and FIH-CTH120-MAD)
  • Plasma PK parameter calculated using a non-compartmental model: tmax (h).

SECONDARY OUTCOMES:
Observed maximum concentration (Cmax). | FIH-CTH120-SAD: On Day 1; FIH-CTH120-MAD: on Day 1, and Day 7
  Secondary Pharmacokinetics endpoints for FIH-CTH120-SAD and FIH-CTH120-MAD (Not applicable for FIH-CTH120-FI).
  • Plasma PK parameter calculated using a non-compartmental model: Cmax (ng/mL).
Observed minimum concentration (Cmin). | FIH-CTH120-SAD: On Day 2; FIH-CTH120-MAD: from Day 2 to Day 7 pre-dose and regularly after the last dose; FIH-CTH120-FI: on Day 2 of Period 1 and Day 15/22/29 of Period 2
  Secondary Pharmacokinetics endpoints for FIH-CTH120-SAD, FIH-CTH120-MAD and FIH-CTH120-FI.
  • Plasma PK parameter calculated using a non-compartmental model: Cmin (ng/mL).
Time to observed maximum concentration (tmax). | FIH-CTH120-SAD: On Day 1; FIH-CTH120-MAD: on Day 1, and Day 7
  Secondary Pharmacokinetics endpoints for FIH-CTH120-SAD and FIH-CTH120-MAD (Not applicable for FIH-CTH120-FI).
  • Plasma PK parameter calculated using a non-compartmental model: tmax (h).
Time to first measurable plasma concentration (tlag). | FIH-CTH120-SAD: On Day 1; FIH-CTH120-MAD: on Day 1, and Day 7; FIH-CTH120-FI: on Day 1 of Period 1 and on Day 14/21/25 of Period 2
  Secondary Pharmacokinetics endpoints for FIH-CTH120-SAD, FIH-CTH120-MAD and FIH-CTH120-FI.
  • Plasma PK parameter calculated using a non-compartmental model: tlag (h).
Time to last measurable plasma concentration (tlast). | FIH-CTH120-SAD: On Day 2; FIH-CTH120-MAD: on Day 1, and Day 7; FIH-CTH120-FI: on Day 2 of Period 1 and Day 15/22/29 of Period 2
  Secondary Pharmacokinetics endpoints for FIH-CTH120-SAD, FIH-CTH120-MAD, and FIH-CTH120-FI.
  • Plasma PK parameter calculated using a non-compartmental model: tlast (h).
Area under the concentration-time curve (AUC0-24h, AUC0-t, AUC0-∞). | FIH-CTH120-SAD: AUC0-24h on Day 1; AUC0-t, AUC0-∞ where t is Day 8 (+/- 1 days) or the latest timepoint observed; FIH-CTH120-MAD: "AUC0-24h on Day 1 and Day 7; AUC0-t, AUC0-∞ after last dose, where t is Day 15 (+ 2 days) or the last timepoint observed
  Secondary Pharmacokinetics endpoints for FIH-CTH120-SAD and FIH-CTH120-MAD (Not applicable for FIH-CTH120-FI).
  • Plasma PK parameter calculated using a non-compartmental model: AUC0-24h (h * ng/mL), AUC0-t (h * ng/mL) AUC0-∞ (h * ng/mL).
Terminal elimination half-life (t1/2). | FIH-CTH120-SAD: from Day 1 to Day 8; FIH-CTH120-MAD: from Day 1 to Day 15; FIH-CTH120-FI: from Day 1 to Day28/35/42
  Secondary Pharmacokinetics endpoints for FIH-CTH120-SAD, FIH-CTH120-MAD, and FIH-CTH120-FI.
  • Plasma PK parameter calculated using a non-compartmental model: t1/2 (h).
Apparent clearance (CL/F). | FIH-CTH120-SAD: from Day 1 to Day 8; FIH-CTH120-MAD: from Day 1 to Day 15; FIH-CTH120-FI: from Day 1 to Day28/35/42
  Secondary Pharmacokinetics endpoints for FIH-CTH120-SAD, FIH-CTH120-MAD, and FIH-CTH120-FI.
  • Plasma PK parameter calculated using a non-compartmental model: CL/F (mL/h * kg).
Apparent volume of distribution: Vd/F. | FIH-CTH120-SAD: from Day 1 to Day 8; FIH-CTH120-MAD: from Day 1 to Day 15; FIH-CTH120-FI: from Day 1 to Day28/35/42
  Secondary Pharmacokinetics endpoints for FIH-CTH120-SAD, FIH-CTH120-MAD, and FIH-CTH120-FI.
  • Plasma PK parameter calculated using a non-compartmental model: Vd/F (mL/kg).
Elimination rate constant (λz). | FIH-CTH120-SAD: from Day 1 to Day 8; FIH-CTH120-MAD: from Day 1 to Day 15; FIH-CTH120-FI: from Day 1 to Day28/35/42
  Secondary Pharmacokinetics endpoints for FIH-CTH120-SAD, FIH-CTH120-MAD, and FIH-CTH120-FI.
  • Plasma PK parameter calculated using a non-compartmental model: λz (1/h).
Serotonin (5-HT) metabolite profile. | FIH-CTH120-SAD: on Day 1 and Day 2; FIH-CTH120-MAD: on Day 1, Day 2, Day 7, and Day 8
  Secondary Pharmacodynamic endpoints for FIH-CTH120-SAD and FIH-CTH120-MAD (Not applicable for FIH-CTH120-FI).
  Concentrations of 5-Hydroxy indoleacetic acid (5-HIAA) (ng/mL).
Noradrenaline (NA) metabolite profile. | FIH-CTH120-SAD: on Day 1 and Day 2; FIH-CTH120-MAD: on Day 1, Day 2, Day 7, and Day 8
  Secondary Pharmacodynamic endpoints for FIH-CTH120-SAD and FIH-CTH120-MAD (Not applicable for FIH-CTH120-FI).
  Concentrations of 3-Methoxy-4-hydroxyphenylglycol (MHPG) (ng/mL).
Treatment-emergent AEs (TAES). | FIH-CTH120-FI: from Day 1 to End-of-study. EOS will be on Day 28, or 35 or 42 (±1 day) depending on the length of the washout period determined
  Secondary Safety and tolerability endpoints (FIH-CTH120-FI).
  • AEs will be described in terms of result, frequency, intensity, medical decision, relation with study drug, as well as treatment received and subject retirement, duration, and time elapsed. AEs will also be listed and coded using the MedDRA Dictionary (version 26.0) for the term's codification.
Treatment-emergent PSCAs in vital signs: blood pressure (mmHg) | FIH-CTH120-FI: from Day 1 to End-of-study. EOS will be on Day 28, or 35 or 42 (±1 day) depending on the length of the washout period determined
  Secondary Safety and tolerability endpoints (FIH-CTH120-FI).
  • Blood pressure (mmHg) will be measured in the supine position following a 5 min rest.
Treatment-emergent PSCAs in vital signs: pulse rate (bpm) | FIH-CTH120-FI: from Day 1 to End-of-study. EOS will be on Day 28, or 35 or 42 (±1 day) depending on the length of the washout period determined
  Secondary Safety and tolerability endpoints (FIH-CTH120-FI).
  • Pulse rate (bpm) will be measured in the supine position following a 5 min rest.
Treatment-emergent PSCAs in vital signs: Oral body temperature (ºC) | FIH-CTH120-FI: from Day 1 to End-of-study. EOS will be on Day 28, or 35 or 42 (±1 day) depending on the length of the washout period determined
  Secondary Safety and tolerability endpoints (FIH-CTH120-FI).
  • Oral body temperature (ºC) will be measured using an automated vital sign monitor device.
Treatment-emergent PSCAs in ECG values: normal sinus rhythm (NSR) | FIH-CTH120-FI: from Day 1 to End-of-study. EOS will be on Day 28, or 35 or 42 (±1 day) depending on the length of the washout period determined
  Secondary Safety and tolerability endpoints (FIH-CTH120-FI).
  • Computerized 12-lead electrocardiogram (ECG) recordings will be obtained. Each lead shall be recorded for at least 3 beats at a speed of 25 mm/s. Triplicate recordings will be made at the time points evaluated. The following parameter will be recorded: normal sinus rhythm (NSR).
Treatment-emergent PSCAs in ECG values: heart rate (bpm) | FIH-CTH120-FI: from Day 1 to End-of-study. EOS will be on Day 28, or 35 or 42 (±1 day) depending on the length of the washout period determined
  Secondary Safety and tolerability endpoints (FIH-CTH120-FI).
  • Computerized 12-lead electrocardiogram (ECG) recordings will be obtained. Each lead shall be recorded for at least 3 beats at a speed of 25 mm/s. Triplicate recordings will be made at the time points evaluated. The following parameters will be recorded: heart rate (bpm).
Treatment-emergent PSCAs in ECG values: PR interval (ms) | FIH-CTH120-FI: from Day 1 to End-of-study. EOS will be on Day 28, or 35 or 42 (±1 day) depending on the length of the washout period determined
  Secondary Safety and tolerability endpoints (FIH-CTH120-FI).
  • Computerized 12-lead electrocardiogram (ECG) recordings will be obtained. Each lead shall be recorded for at least 3 beats at a speed of 25 mm/s. Triplicate recordings will be made at the time points evaluated. The following parameter will be recorded: PR interval (ms)
Treatment-emergent PSCAs in ECG values: QRS duration (ms) | FIH-CTH120-FI: from Day 1 to End-of-study. EOS will be on Day 28, or 35 or 42 (±1 day) depending on the length of the washout period determined
  Secondary Safety and tolerability endpoints (FIH-CTH120-FI).
  • Computerized 12-lead electrocardiogram (ECG) recordings will be obtained. Each lead shall be recorded for at least 3 beats at a speed of 25 mm/s. Triplicate recordings will be made at the time points evaluated. The following parameter will be recorded: QRS duration (ms).
Treatment-emergent PSCAs in ECG values: QT (ms) | FIH-CTH120-FI: from Day 1 to End-of-study. EOS will be on Day 28, or 35 or 42 (±1 day) depending on the length of the washout period determined
  Secondary Safety and tolerability endpoints (FIH-CTH120-FI).
  • Computerized 12-lead electrocardiogram (ECG) recordings will be obtained. Each lead shall be recorded for at least 3 beats at a speed of 25 mm/s. Triplicate recordings will be made at the time points evaluated. The following parameter will be recorded: QT (ms).
Treatment-emergent PSCAs in ECG values: QTcF (ms) | FIH-CTH120-FI: from Day 1 to End-of-study. EOS will be on Day 28, or 35 or 42 (±1 day) depending on the length of the washout period determined
  Secondary Safety and tolerability endpoints (FIH-CTH120-FI).
  • Computerized 12-lead electrocardiogram (ECG) recordings will be obtained. Each lead shall be recorded for at least 3 beats at a speed of 25 mm/s. Triplicate recordings will be made at the time points evaluated. The following parameter will be recorded: QTcF (ms).
Treatment-emergent PSCAs in safety laboratory parameters: haematology | FIH-CTH120-FI: from Day 1 to End-of-study. EOS will be on Day 28, or 35 or 42 (±1 day) depending on the length of the washout period determined
  Secondary Safety and tolerability endpoints (FIH-CTH120-FI). The following tests will be performed:
  • Haematology: complete blood count (complete blood count [CBC]; including haemoglobin, haematocrit, red blood cell [RBC], white blood cell (WBC), platelet count, and percent and absolute differential count (neutrophils, lymphocytes, eosinophils, monocytes, basophils, and other cells).
Treatment-emergent PSCAs in safety laboratory parameters: serum chemistry | FIH-CTH120-FI: from Day 1 to End-of-study. EOS will be on Day 28, or 35 or 42 (±1 day) depending on the length of the washout period determined
  Secondary Safety and tolerability endpoints (FIH-CTH120-FI). The following tests will be performed:
  • Serum chemistry: sodium, potassium, chloride, non-fasting glucose, urea, creatinine, calcium, phosphate, magnesium, total and direct bilirubin, total protein, albumin, ALT, AST, ALP, lactate dehydrogenase.
Treatment-emergent PSCAs in safety laboratory parameters: coagulation | FIH-CTH120-FI: from Day 1 to End-of-study. EOS will be on Day 28, or 35 or 42 (±1 day) depending on the length of the washout period determined
  Secondary Safety and tolerability endpoints (FIH-CTH120-FI). The following tests will be performed:
  • Coagulation parameters: activated partial thromboplastin time (aPTT), PT and INR.
Treatment-emergent PSCAs in safety laboratory parameters: urinalysis | FIH-CTH120-FI: from Day 1 to End-of-study. EOS will be on Day 28, or 35 or 42 (±1 day) depending on the length of the washout period determined
  Secondary Safety and tolerability endpoints (FIH-CTH120-FI). The following tests will be performed:
  • Urinalysis parameters:
  * Macroscopic examination: specific gravity, pH, protein, glucose, ketones, blood, bilirubin, leukocyte, urobilinogen, and nitrite.
  * Microscopic examination: RBCs, WBCs, epithelial cells, casts, crystals, bacteria, and yeast.
Psychometric tests: HADS | FIH-CTH120-FI: On Day -1, Day 2, Day 13/20/27 and Day 15/22/29
  Secondary Safety and tolerability endpoints (FIH-CTH120-FI).
  • HADS: Self-reported questionnaire used to detect depression and anxiety. It consists of 14 items (7 related to depression and 7 to anxiety) scored using a 4-point Likert scale (each item ranging from 0 to 3). Two scores are generated one for depression and one for anxiety ranging each score ranging from 0 to 21. Higher scores indicate greater levels of anxiety or depression. Both scores can be categorized into: Normality (0-7); Probable case of anxiety or depression (8-10); Case of anxiety or depression (11-21).
Psychometric tests: IMS | FIH-CTH120-FI: On Day -1, Day 2, Day 13/20/27 and Day 15/22/29
  Secondary Safety and tolerability endpoints (FIH-CTH120-FI).
  • IMS: The IMS is a tool to remotely and quickly track mood changes related to depression and anxiety in the moment. It consists of 22 items, scored between 1 and 7. The total score for this scale is the sum of the scores on all 22 items: ranging from 22 to 154. Lower scores reflect more negative mood states.

OTHER OUTCOMES:
Area under the concentration-time curve (AUC0-24h, AUC0-t, AUC0-∞). | FIH-CTH120-FI: AUC0-24h on Day 1; AUC0-t, AUC0-∞ where t is the last or the latest timepoint observed
  Exploratory objective (FIH-CTH120-FI). Plasma pharmacokinetics of the major metabolite of CTH120 after CTH120 single dose administration.
  • Plasma PK parameter calculated using a non-compartmental model: AUC0-24h (h * ng/mL), AUC0-t (h * ng/mL) AUC0-∞ (h * ng/mL).
Observed maximum concentration (Cmax). | FIH-CTH120-FI: on Day 1 of Period 1 and on Day 14/21/25 of Period 2
  Exploratory objective (FIH-CTH120-FI). Plasma pharmacokinetics of the major metabolite of CTH120 after CTH120 single dose administration.
  • Plasma PK parameter calculated using a non-compartmental model: Cmax (ng/mL).
Time to observed maximum concentration (tmax). | FIH-CTH120-FI: on Day 1 of Period 1 and on Day 14/21/25 of Period 2
  Exploratory objective (FIH-CTH120-FI). Plasma pharmacokinetics of the major metabolite of CTH120 after CTH120 single dose administration.
  • Plasma PK parameter calculated using a non-compartmental model: tmax (h).
Observed minimum concentration (Cmin). | FIH-CTH120-FI: on Day 2 of Period 1 and Day 15/22/29 of Period 2
  Exploratory objective (FIH-CTH120-FI). Plasma pharmacokinetics of the major metabolite of CTH120 after CTH120 single dose administration.
  • Plasma PK parameter calculated using a non-compartmental model: Cmin (ng/mL).
Time to first measurable plasma concentration (tlag). | FIH-CTH120-FI: on Day 1 of Period 1 and on Day 14/21/25 of Period 2
  Exploratory objective (FIH-CTH120-FI). Plasma pharmacokinetics of the major metabolite of CTH120 after CTH120 single dose administration.
  • Plasma PK parameter calculated using a non-compartmental model: tlag (h).
Time to last measurable plasma concentration (tlast). | FIH-CTH120-FI: on Day 2 of Period 1 and Day 15/22/29 of Period 2
  Exploratory objective (FIH-CTH120-FI). Plasma pharmacokinetics of the major metabolite of CTH120 after CTH120 single dose administration.
  • Plasma PK parameter calculated using a non-compartmental model: tlast (h).
Terminal elimination half-life (t1/2). | FIH-CTH120-FI: from Day 1 to Day28/35/42
  Exploratory objective (FIH-CTH120-FI).
  • Plasma PK parameter calculated using a non-compartmental model: t1/2 (h).
Metabolic ratio Cmax (MR Cmax) | FIH-CTH120-FI: from Day 1 to Day28/35/42
  Exploratory objective (FIH-CTH120-FI). Plasma pharmacokinetics of the major metabolite of CTH120 after CTH120 single dose administration.
  • Plasma PK parameter calculated using a non-compartmental model: MR Cmax (n-fold).
Metabolic ratio AUC0-24 (MR AUC0-24) | FIH-CTH120-FI: from Day 1 to Day28/35/42
  Exploratory objective (FIH-CTH120-FI). Plasma pharmacokinetics of the major metabolite of CTH120 after CTH120 single dose administration.
  • Plasma PK parameter calculated using a non-compartmental model: MR AUC0-24 (n-fold)
Elimination rate constant (λz) | FIH-CTH120-FI: from Day 1 to Day28/35/42
  Exploratory objective (FIH-CTH120-FI). Plasma pharmacokinetics of the major metabolite of CTH120 after CTH120 single dose administration.
  • Plasma PK parameter calculated using a non-compartmental model: λz (1/h).
Renal clearance (CLr) | FIH-CTH120-FI: from Day 1 to Day28/35/42
  Exploratory objective (FIH-CTH120-FI). Urine pharmacokinetics of the major metabolite of CTH120 after CTH120 single dose administration.
  Renal clearance (L/h), as a Volume/time, calculated as CLr = Ae/PlasmaAUC0-∞, where Ae (µg) is the cumulative amount of unchanged drug excreted into the urine (0-48 h interval) and Plasma AUC0-∞ (ng.h/mL) is the area under the plasma concentration-time curve from time zero to infinity.
Amount excreted: absolute value as Ae | FIH-CTH120-FI: from Day 1 to Day28/35/42
  Exploratory objective (FIH-CTH120-FI). Urine pharmacokinetics of the major metabolite of CTH120 after CTH120 single dose administration.
  • The excreted amount will be calculated as absolute value as Ae: cumulative amount of unchanged drug excreted into the urine (interval) (µg).
Amount excreted: relative to dose as fe/F | FIH-CTH120-FI: from Day 1 to Day28/35/42
  Exploratory objective (FIH-CTH120-FI). Urine pharmacokinetics of the major metabolite of CTH120 after CTH120 single dose administration.
  • The excreted amount will be calculated as relative to dose as fe/F: fraction of the oral administered drug excreted into the urine (%).
Urinary excretion rate (UER) | FIH-CTH120-FI: from Day 1 to Day28/35/42
  Exploratory objective (FIH-CTH120-FI). Urine pharmacokinetics of the major metabolite of CTH120 after CTH120 single dose administration.
  The urinary excretion rate (μg/h) is the product of the urine flow rate (mL/h) and the urine analyte concentration (ng/mL), where:
  * Urine flow rate (UFR) is the quotient between the Urine volume (mL) and the time interval (h), where urine volume is the total urine volume collected in the time interval (mL).
  * Urine analyte concentration: concentration of the analyte in urine (ng/mL).
Urine elimination rate constant (h-1) | FIH-CTH120-FI: from Day 1 to Day28/35/42
  Exploratory objective (FIH-CTH120-FI). Urine pharmacokinetics of the major metabolite of CTH120 after CTH120 single dose administration.
  • Urine elimination rate constant (h-1): calculated as the slope (semilog plot) of the cumulative amount of drug excreted after each collection interval against the median of the collection interval. Nominal or actual times can be used as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael De la Torre, Pharm, PhD, Principal Investigator — Hospital del Mar Medical Research Institute (IMIM)
Locations (1):
- Hospital del Mar Medical Research Institute (IMIM), Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Myrick LK, Nakamoto-Kinoshita M, Lindor NM, Kirmani S, Cheng X, Warren ST. Fragile X syndrome due to a missense mutation. Eur J Hum Genet. 2014 Oct;22(10):1185-9. doi: 10.1038/ejhg.2013.311. Epub 2014 Jan 22. PMID 24448548
- [Background] Quartier A, Poquet H, Gilbert-Dussardier B, Rossi M, Casteleyn AS, Portes VD, Feger C, Nourisson E, Kuentz P, Redin C, Thevenon J, Mosca-Boidron AL, Callier P, Muller J, Lesca G, Huet F, Geoffroy V, El Chehadeh S, Jung M, Trojak B, Le Gras S, Lehalle D, Jost B, Maury S, Masurel A, Edery P, Thauvin-Robinet C, Gerard B, Mandel JL, Faivre L, Piton A. Intragenic FMR1 disease-causing variants: a significant mutational mechanism leading to Fragile-X syndrome. Eur J Hum Genet. 2017 Apr;25(4):423-431. doi: 10.1038/ejhg.2016.204. Epub 2017 Feb 8. PMID 28176767
- [Background] Hagerman RJ, Berry-Kravis E, Hazlett HC, Bailey DB Jr, Moine H, Kooy RF, Tassone F, Gantois I, Sonenberg N, Mandel JL, Hagerman PJ. Fragile X syndrome. Nat Rev Dis Primers. 2017 Sep 29;3:17065. doi: 10.1038/nrdp.2017.65. PMID 28960184
- [Background] Wang LW, Berry-Kravis E, Hagerman RJ. Fragile X: leading the way for targeted treatments in autism. Neurotherapeutics. 2010 Jul;7(3):264-74. doi: 10.1016/j.nurt.2010.05.005. PMID 20643379
- [Background] Grigsby J. The fragile X mental retardation 1 gene (FMR1): historical perspective, phenotypes, mechanism, pathology, and epidemiology. Clin Neuropsychol. 2016 Aug;30(6):815-33. doi: 10.1080/13854046.2016.1184652. Epub 2016 Jun 29. PMID 27356167
- [Background] Banerjee A, Ifrim MF, Valdez AN, Raj N, Bassell GJ. Aberrant RNA translation in fragile X syndrome: From FMRP mechanisms to emerging therapeutic strategies. Brain Res. 2018 Aug 15;1693(Pt A):24-36. doi: 10.1016/j.brainres.2018.04.008. Epub 2018 Apr 10. PMID 29653083
- [Background] Bakker CE, Oostra BA. Understanding fragile X syndrome: insights from animal models. Cytogenet Genome Res. 2003;100(1-4):111-23. doi: 10.1159/000072845. PMID 14526171
- [Background] Darnell JC, Klann E. The translation of translational control by FMRP: therapeutic targets for FXS. Nat Neurosci. 2013 Nov;16(11):1530-6. doi: 10.1038/nn.3379. Epub 2013 Apr 14. PMID 23584741
- [Background] Richter JD, Bassell GJ, Klann E. Dysregulation and restoration of translational homeostasis in fragile X syndrome. Nat Rev Neurosci. 2015 Oct;16(10):595-605. doi: 10.1038/nrn4001. Epub 2015 Sep 9. PMID 26350240
- [Background] Gholizadeh S, Halder SK, Hampson DR. Expression of fragile X mental retardation protein in neurons and glia of the developing and adult mouse brain. Brain Res. 2015 Jan 30;1596:22-30. doi: 10.1016/j.brainres.2014.11.023. Epub 2014 Nov 20. PMID 25446451
- [Background] Feng Y, Gutekunst CA, Eberhart DE, Yi H, Warren ST, Hersch SM. Fragile X mental retardation protein: nucleocytoplasmic shuttling and association with somatodendritic ribosomes. J Neurosci. 1997 Mar 1;17(5):1539-47. doi: 10.1523/JNEUROSCI.17-05-01539.1997. PMID 9030614
- [Background] Hanson AC, Hagerman RJ. Serotonin dysregulation in Fragile X Syndrome: implications for treatment. Intractable Rare Dis Res. 2014 Nov;3(4):110-7. doi: 10.5582/irdr.2014.01027. PMID 25606361
- [Background] Boccuto L, Chen CF, Pittman AR, Skinner CD, McCartney HJ, Jones K, Bochner BR, Stevenson RE, Schwartz CE. Decreased tryptophan metabolism in patients with autism spectrum disorders. Mol Autism. 2013 Jun 3;4(1):16. doi: 10.1186/2040-2392-4-16. PMID 23731516
- [Background] Chandana SR, Behen ME, Juhasz C, Muzik O, Rothermel RD, Mangner TJ, Chakraborty PK, Chugani HT, Chugani DC. Significance of abnormalities in developmental trajectory and asymmetry of cortical serotonin synthesis in autism. Int J Dev Neurosci. 2005 Apr-May;23(2-3):171-82. doi: 10.1016/j.ijdevneu.2004.08.002. PMID 15749243
- [Background] Wang H, Wu LJ, Kim SS, Lee FJ, Gong B, Toyoda H, Ren M, Shang YZ, Xu H, Liu F, Zhao MG, Zhuo M. FMRP acts as a key messenger for dopamine modulation in the forebrain. Neuron. 2008 Aug 28;59(4):634-47. doi: 10.1016/j.neuron.2008.06.027. PMID 18760699
- [Background] Gkogkas CG, Khoutorsky A, Cao R, Jafarnejad SM, Prager-Khoutorsky M, Giannakas N, Kaminari A, Fragkouli A, Nader K, Price TJ, Konicek BW, Graff JR, Tzinia AK, Lacaille JC, Sonenberg N. Pharmacogenetic inhibition of eIF4E-dependent Mmp9 mRNA translation reverses fragile X syndrome-like phenotypes. Cell Rep. 2014 Dec 11;9(5):1742-1755. doi: 10.1016/j.celrep.2014.10.064. Epub 2014 Nov 26. PMID 25466251
- [Background] Wahlstrom-Helgren S, Klyachko VA. GABAB receptor-mediated feed-forward circuit dysfunction in the mouse model of fragile X syndrome. J Physiol. 2015 Nov 15;593(22):5009-24. doi: 10.1113/JP271190. Epub 2015 Oct 2. PMID 26282581
- [Background] Kashima R, Roy S, Ascano M, Martinez-Cerdeno V, Ariza-Torres J, Kim S, Louie J, Lu Y, Leyton P, Bloch KD, Kornberg TB, Hagerman PJ, Hagerman R, Lagna G, Hata A. Augmented noncanonical BMP type II receptor signaling mediates the synaptic abnormality of fragile X syndrome. Sci Signal. 2016 Jun 7;9(431):ra58. doi: 10.1126/scisignal.aaf6060. PMID 27273096
- [Background] Sidhu H, Dansie LE, Hickmott PW, Ethell DW, Ethell IM. Genetic removal of matrix metalloproteinase 9 rescues the symptoms of fragile X syndrome in a mouse model. J Neurosci. 2014 Jul 23;34(30):9867-79. doi: 10.1523/JNEUROSCI.1162-14.2014. PMID 25057190
- [Background] Pasciuto E, Ahmed T, Wahle T, Gardoni F, D'Andrea L, Pacini L, Jacquemont S, Tassone F, Balschun D, Dotti CG, Callaerts-Vegh Z, D'Hooge R, Muller UC, Di Luca M, De Strooper B, Bagni C. Dysregulated ADAM10-Mediated Processing of APP during a Critical Time Window Leads to Synaptic Deficits in Fragile X Syndrome. Neuron. 2015 Jul 15;87(2):382-98. doi: 10.1016/j.neuron.2015.06.032. PMID 26182420
- [Background] Danesi C, Achuta VS, Corcoran P, Peteri UK, Turconi G, Matsui N, Albayrak I, Rezov V, Isaksson A, Castren ML. Increased Calcium Influx through L-type Calcium Channels in Human and Mouse Neural Progenitors Lacking Fragile X Mental Retardation Protein. Stem Cell Reports. 2018 Dec 11;11(6):1449-1461. doi: 10.1016/j.stemcr.2018.11.003. Epub 2018 Nov 29. PMID 30503263
- [Background] Pilaz LJ, Lennox AL, Rouanet JP, Silver DL. Dynamic mRNA Transport and Local Translation in Radial Glial Progenitors of the Developing Brain. Curr Biol. 2016 Dec 19;26(24):3383-3392. doi: 10.1016/j.cub.2016.10.040. Epub 2016 Dec 1. PMID 27916527
- [Background] Bailey DB Jr, Raspa M, Olmsted M, Holiday DB. Co-occurring conditions associated with FMR1 gene variations: findings from a national parent survey. Am J Med Genet A. 2008 Aug 15;146A(16):2060-9. doi: 10.1002/ajmg.a.32439. PMID 18570292
- [Background] Berry-Kravis E, Raspa M, Loggin-Hester L, Bishop E, Holiday D, Bailey DB. Seizures in fragile X syndrome: characteristics and comorbid diagnoses. Am J Intellect Dev Disabil. 2010 Nov;115(6):461-72. doi: 10.1352/1944-7558-115.6.461. PMID 20945999
- [Background] McLennan Y, Polussa J, Tassone F, Hagerman R. Fragile x syndrome. Curr Genomics. 2011 May;12(3):216-24. doi: 10.2174/138920211795677886. PMID 22043169
- [Background] Sauna-Aho O, Bjelogrlic-Laakso N, Siren A, Arvio M. Signs indicating dementia in Down, Williams and Fragile X syndromes. Mol Genet Genomic Med. 2018 Sep;6(5):855-860. doi: 10.1002/mgg3.430. Epub 2018 Jul 3. PMID 29971948
- [Background] Bartholomay KL, Lee CH, Bruno JL, Lightbody AA, Reiss AL. Closing the Gender Gap in Fragile X Syndrome: Review on Females with FXS and Preliminary Research Findings. Brain Sci. 2019 Jan 12;9(1):11. doi: 10.3390/brainsci9010011. PMID 30642066
- [Background] Cordeiro L, Ballinger E, Hagerman R, Hessl D. Clinical assessment of DSM-IV anxiety disorders in fragile X syndrome: prevalence and characterization. J Neurodev Disord. 2011 Mar;3(1):57-67. doi: 10.1007/s11689-010-9067-y. Epub 2010 Dec 3. PMID 21475730
- [Background] Utari A, Adams E, Berry-Kravis E, Chavez A, Scaggs F, Ngotran L, Boyd A, Hessl D, Gane LW, Tassone F, Tartaglia N, Leehey MA, Hagerman RJ. Aging in fragile X syndrome. J Neurodev Disord. 2010 Jun;2(2):70-76. doi: 10.1007/s11689-010-9047-2. Epub 2010 May 12. PMID 20585378
- [Background] Tassone F. Advanced technologies for the molecular diagnosis of fragile X syndrome. Expert Rev Mol Diagn. 2015;15(11):1465-73. doi: 10.1586/14737159.2015.1101348. Epub 2015 Oct 21. PMID 26489042
- [Background] Rajan-Babu IS, Chong SS. Molecular Correlates and Recent Advancements in the Diagnosis and Screening of FMR1-Related Disorders. Genes (Basel). 2016 Oct 14;7(10):87. doi: 10.3390/genes7100087. PMID 27754417
- [Background] Kidd SA, Lachiewicz A, Barbouth D, Blitz RK, Delahunty C, McBrien D, Visootsak J, Berry-Kravis E. Fragile X syndrome: a review of associated medical problems. Pediatrics. 2014 Nov;134(5):995-1005. doi: 10.1542/peds.2013-4301. Epub 2014 Oct 6. PMID 25287458
- [Background] Crawford DC, Acuna JM, Sherman SL. FMR1 and the fragile X syndrome: human genome epidemiology review. Genet Med. 2001 Sep-Oct;3(5):359-71. doi: 10.1097/00125817-200109000-00006. PMID 11545690
- [Background] Tassone F, Iong KP, Tong TH, Lo J, Gane LW, Berry-Kravis E, Nguyen D, Mu LY, Laffin J, Bailey DB, Hagerman RJ. FMR1 CGG allele size and prevalence ascertained through newborn screening in the United States. Genome Med. 2012 Dec 21;4(12):100. doi: 10.1186/gm401. eCollection 2012. PMID 23259642
- [Background] Hunter J, Rivero-Arias O, Angelov A, Kim E, Fotheringham I, Leal J. Epidemiology of fragile X syndrome: a systematic review and meta-analysis. Am J Med Genet A. 2014 Jul;164A(7):1648-58. doi: 10.1002/ajmg.a.36511. Epub 2014 Apr 3. PMID 24700618
- [Background] Coffee B, Keith K, Albizua I, Malone T, Mowrey J, Sherman SL, Warren ST. Incidence of fragile X syndrome by newborn screening for methylated FMR1 DNA. Am J Hum Genet. 2009 Oct;85(4):503-14. doi: 10.1016/j.ajhg.2009.09.007. PMID 19804849
- [Background] Sibille M, Patat A, Caplain H, Donazzolo Y. A safety grading scale to support dose escalation and define stopping rules for healthy subject first-entry-into-man studies: some points to consider from the French Club Phase I working group. Br J Clin Pharmacol. 2010 Nov;70(5):736-48. doi: 10.1111/j.1365-2125.2010.03741.x. PMID 21039768
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Herrero MJ, Blanch J, Peri JM, De Pablo J, Pintor L, Bulbena A. A validation study of the hospital anxiety and depression scale (HADS) in a Spanish population. Gen Hosp Psychiatry. 2003 Jul-Aug;25(4):277-83. doi: 10.1016/s0163-8343(03)00043-4. PMID 12850660
- [Background] Nahum M, Van Vleet TM, Sohal VS, Mirzabekov JJ, Rao VR, Wallace DL, Lee MB, Dawes H, Stark-Inbar A, Jordan JT, Biagianti B, Merzenich M, Chang EF. Immediate Mood Scaler: Tracking Symptoms of Depression and Anxiety Using a Novel Mobile Mood Scale. JMIR Mhealth Uhealth. 2017 Apr 12;5(4):e44. doi: 10.2196/mhealth.6544. PMID 28404542
- See also: EMEA, "Committee for Medicinal Products for Human Use (CHMP) Guideline on strategies to identify and mitigate risks for first-in-human and early clinical trials with investigational medicinal products," EMEA/CHMP/SWP/28367/07, 2017 — https://www.ema.europa.eu/en/documents/scientific-guideline/guideline-strategies-identify-mitigate-risks-first-human-early-clinical-trials-investigational_en.pdf
- See also: FDA, Guidance for Industry Estimating the Maximum Safe Starting Dose in Initial Clinical Trials for Therapeutics in Adult Healthy Volunteers Pharmacology and Toxicology Guidance for Industry..... — https://www.fda.gov/media/72309/download
- See also: FDA, "Assessment of Abuse Potential of Drugs Guidance for Industry," 2017, Accessed: Jul. 07, 2022. — https://www.fda.gov/media/116739/download
- See also: FDA, "FDA Guidance for Industry Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials - ECA Academy." — https://www.gmp-compliance.org/guidelines/gmp-guideline/fda-guidance-for-industrytoxicity-grading-scale-for-healthy-adult-and-adolescent-volunteers-enrolled-in-preventive-vaccine-clini
- See also: "FDA Guidance for Industry: Food-Effect Bioavailability and Fed Bioequivalence Studies (Issued 12/2002, Posted 1/30/2003) - ECA Academy." — https://www.gmp-compliance.org/guidelines/gmp-guideline/fda-guidance-for-industry-food-effect-bioavailability-and-fed-bioequivalence-studies-issued-12-2002-posted-1-30-2003
- See also: U.S. DEPARTMENT OF HEALTH AND HUMAN SERVICES, "Common Terminology Criteria for Adverse Events (CTCAE) v5.0," 2017 — https://ctep.cancer.gov/protocoldevelopment/electronic_applications/ctc.htm
- See also: N. Cancer Institute, "Common Terminology Criteria for Adverse Events (CTCAE) Common Terminology Criteria for Adverse Events (CTCAE) v5.0," 2017 — https://ctep.cancer.gov/protocoldevelopment/electronic_applications/ctc.htm